CLINICAL TRIAL: NCT02156440
Title: A Double Blind, Placebo Controlled Cross Over Study to Explore the Efficacy of SierraSil® Joint Formula 14™ in Adults With Osteoarthritis of the Knee
Brief Title: Cross-over Study of the Efficacy and Safety of SierraSil Joint Formula 14 in Osteoarthritis of the Knee
Acronym: 11SOHS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: SierraSil Health Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 11SOHS
Record Dates: First submitted 2014-06-02; First posted 2014-06-05 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Osteoarthritis of the Knee
Keywords: Ostearthritis; Knee; SierraSil
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsules: one capsule taken 3 times per day with water. Subjects are to drink 6 to 8 glasses of water daily.
  Interventions: Dietary Supplement: Placebo
- SierraSil Joint Formula 14 (Experimental): SierraSil Joint Formula 14 capsules: one capsule taken 3 times per day with water. Subjects are to drink 6 to 8 glasses of water daily.
  Interventions: Dietary Supplement: SierraSil Joint Formula 14

INTERVENTIONS:
Dietary Supplement: SierraSil Joint Formula 14 — 667 mg SierraSil® hydrothermal mineral complex
  Other Names: SierraSil® hydrothermal mineral complex
  Arms: SierraSil Joint Formula 14
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
Osteoarthritis (OA) affects approximately 10% of people older than 60 years, and compromises the quality of life of more than 21 million North Americans. Studies on the use of complimentary and alternative medicines have reported that OA patients in the US are among the highest users of CAM. Previous studies on a unique natural mineral product SierraSil® demonstrated an improvement in joint health and function in subjects with mild to moderate OA of the knee. Extracts of Sierrasil® are reported to reduce cartilage degradation in response to IL-8 and nitric oxide production suggesting an ability to suppress IL-8 mediated events in human cartilage. The primary objective is to assess the efficacy of SeirraSil Joint Formula versus placebo on the symptoms of osteoarthritis as assessed by WOMAC™ Osteoarthritis Index Pain subscale in subjects with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age
* If female, subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

OR

Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Intrauterine devices
* Vasectomy of partner (shown successful as per appropriate follow-up)
* Abstinence
* Primary or secondary, unilateral or bilateral osteoarthritis of the knee (American College of Rheumatology Clinical Criteria for Classification)

Knee pain with at least 3 of the following:

* Age > 50 years
* Stiffness < 30 minutes
* Crepitus
* Bony Tenderness
* Bony enlargement
* No palpable warmth
* Self reported difficulty performing at least one of the following activities because of knee pain:
* lifting and carrying groceries
* walking one-quarter of a mile
* getting in and out of a chair
* going up and down stairs
* mobility
* self-care activities
* Able to walk unassisted (may use walking stick, crutch, or knee brace)
* Availability for duration of study period (14 weeks)
* Subject using other therapies for OA, such as exercise, heat/cold therapy, joint protection and physiotherapy/occupational therapy agrees to continue these therapies as normal avoiding changes in frequency or intensity and to record therapies in the study diary
* Subject agrees not to start any new therapies for OA during the course of the study
* Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
* Subject has a diagnosis of rheumatoid arthritis, fibromyalgia, spinal disorders or other musculoskeletal disease
* Subject has been recommended for knee surgery
* Subject has hemosiderosis or hemochromatosis
* Subject has kidney or liver disease, blood disorders, active cancer and/or HIV infection
* Subject has significant medical history or current metabolic disorders, thyroid disease, immune disorders and/or cardiovascular disease will be reviewed by the Qualified Investigator (QI). Subjects deemed by the QI to be at possible risk will not be permitted in this study.
* Use of illicit drugs or history of drug or alcohol abuse with the past 5 years (currently having more than 2 standard alcoholic drinks per day)
* Planned surgery during the course of the trial
* Use of intra-articular, oral or parenteral corticosteroids, or other injectable prescription medication (e.g., Synvisc) within 2 months prior to randomization and during the trial
* Requires the use of prescription drugs to control pain (other than provided rescue medication)
* Use of oral or topical prescription or over the counter medications or natural health products for pain relief 48 hours prior to randomization and during the trial (other than provided rescue medication)
* Use of iron supplementation during the trial (i.e. provided by multivitamins, prescription medication, or any other mineral preparations containing iron)
* Use of antacids containing aluminum and other aluminum containing medications or supplements during the trial
* Clinically significant abnormal laboratory results at screening
* Abnormal serum ferritin levels ≥200 µg/L
* Abnormal serum aluminum levels >16 µg/L
* eGFR < 60 and abnormal liver function tests
* Allergy or sensitivity to test product ingredients
* Individuals who are cognitively impaired and/or who are unable to give informed consent
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
WOMAC osteoarthritis index Pain Subscale as a measure of osteoarthritis pain | 4 weeks
  Assessed during each 4 week treatment period

SECONDARY OUTCOMES:
WOMAC osteoarthritis index Stiffness subscale as a measure of osteoarthritis stiffness | 4 weeks
  Assessed during each 4 week treatment period
WOMAC osteoarthritis index Physical Function subscale as a measure of physical function | 4 weeks
  Assessed during each 4 week treatment period
SF-36 questionnaire score as a measure of Quality of Life | 4 weeks
  Assessed during each 4 week treatment period
Inflammatory markers | 4 weeks
  hsCRP, TNF-alpha, IL-6 assessed during each 4 week treatment period
Amount of Rescue Medication Used | 4 weeks
  Assessed during each 4 week treatment period
Vital Signs | 4 weeks
  Blood pressure, heart rate, weight and BMI were assessed during each 4 week treatment period
Safety Blood Parameters | 4 weeks
  CBC, electrolytes, fasting glucose, creatinine, eGFR AST, ALT, GGT, bilirubin, creatine kinase, aluminum, ferritin, TIBC and iron saturation were assessed during each of the 4 week treatment periods
Number of participants with Adverse Events as measure of safety | 4 weeks
  Assessed during each 4 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada